CLINICAL TRIAL: NCT06977633
Title: A pH-Responsive Hydrogel Microneedle Patch for Continuous Measurement of Ketone Bodies and Glucose: CGM-CKM
Brief Title: Feasibility Study of a Continuous Glucose-Ketone Monitoring Device in People With Type 1 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahla Poudineh (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor-Investigator, Mahla Poudineh, Assistant Professor, University of Waterloo
Organization: University of Waterloo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 76354
Record Dates: First submitted 2025-04-18; First posted 2025-05-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes (T1D)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a single-group, non-randomized study designed to evaluate the accuracy of an investigational continuous glucose ketone sensor in participants with type 1 diabetes. Under controlled inpatient conditions, sensor readings will be compared to reference standards for blood glucose and ketone levels. The study does not include therapeutic interventions or real-time clinical decision-making based on sensor output.
Masking Description: No masking will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- People with type 1 diabetes on insulin pump (Experimental)
  Interventions: Behavioral: Temporary Insulin Suspension; Device: Glucose and ketone sensor

INTERVENTIONS:
Behavioral: Temporary Insulin Suspension — Participants will suspend insulin delivery from their personal insulin pumps for up to 3 hours. Insulin suspension is temporary and participant-driven under supervision.
Device: Glucose and ketone sensor — The participants wear a prototype continuous glucose-ketone monitoring (CGM-CKM) device using painless hydrogel microneedles for 4 hours.

SUMMARY:
The goal of this study is to evaluate a CGM-CKM device during insulin suspension in patients with type 1 diabetes. 10 patients with T1D will be recruited for a pilot study. The patients will visit CTRU at Stanford Medical School. The CGM-CKM device will be applied to the upper arm area of patients and baseline ketone and glucose measurement will be performed for one hour prior to suspending or disconnecting the pump. Upon baseline measurement, the pump will be disconnected for 3 hours while the electrochemical signals are collected from the CGM-CKM device. During the 3 hours of pump disconnection, blood samples will be collected every 5 minutes from participants for analyzing their insulin and glucagon using conventional ELISA kits and glucose and ketone using standard meters.

DETAILED DESCRIPTION:
This is a non-significant risk (NSR) device study not conducted under an IDE, in accordance with 21 CFR 812.2(b)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least 1 year without significant endogenous insulin production
* Currently using insulin pump
* Understanding and willingness to follow the protocol and sign informed consent.
* Willingness to sign a consent for release of medical information at the time of enrollment
* Ability to speak, read and write in the language of the investigators.

Exclusion Criteria:

* History of DKA or severe hypoglycemia within the past 6 months
* eGFR <45 mL/min/1.73 m2 or other significant renal impairment
* Pregnancy or breastfeeding
* Current use of non-insulin medications affecting ketone production, including SGLT2 inhibitors
* Active skin infections or conditions affecting sensor application sites
* Known skin allergies to tapes or adhesives
* Current use of any long-acting insulin analogs
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of Glucose Measured by Experimental CGM-CKM Sensor Compared to Blood Glucose | 5 hours
  Correlation between glucose concentrations (mmol/L) measured by the CGM-CKM sensor and plasma glucose concentrations measured with YSI 2300 glucose analyzer.
Concentration of Ketones Measured by Experimental CGM-CKM Sensor Compared to Blood Ketones | 5 hours
  Correlation between ketone concentrations (mmol/L) measured by the experimental CKM-CKM sensor and blood ketone concentrations measured using commercially available tests.

SECONDARY OUTCOMES:
Plasma Insulin Concentration Measured by Mercodia ELISA Assay | 5 hours
  Insulin concentration (pmol/L) in plasma samples collected during the study will be measured using Mercodia insulin ELISA assay.
Plasma Glucagon Concentration Measured by Mercodia ELISA Assay | 5 hours
  Glucagon concentration (pmol/L) in plasma samples collected during the study will be measured using Mercodia insulin ELISA assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Sensor measurements and blood plasma levels will be shared via journal/conference publications.

REFERENCES:
- [Background] Ausri IR, Sadeghzadeh S, Biswas S, Zheng H, GhavamiNejad P, Huynh MDT, Keyvani F, Shirzadi E, Rahman FA, Quadrilatero J, GhavamiNejad A, Poudineh M. Multifunctional Dopamine-Based Hydrogel Microneedle Electrode for Continuous Ketone Sensing. Adv Mater. 2024 Aug;36(32):e2402009. doi: 10.1002/adma.202402009. Epub 2024 Jun 16. PMID 38847967
- [Background] GhavamiNejad P, GhavamiNejad A, Zheng H, Dhingra K, Samarikhalaj M, Poudineh M. A Conductive Hydrogel Microneedle-Based Assay Integrating PEDOT:PSS and Ag-Pt Nanoparticles for Real-Time, Enzyme-Less, and Electrochemical Sensing of Glucose. Adv Healthc Mater. 2023 Jan;12(1):e2202362. doi: 10.1002/adhm.202202362. Epub 2022 Oct 13. PMID 36183355